CLINICAL TRIAL: NCT05505045
Title: Feasibility of Using Remotely-delivered Metacognitive Strategy Training to Address Cancer-related Cognitive Impairment in Breast Cancer
Brief Title: Metacognitive Strategy Training in Cancer-related Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Anna Boone, Assistant Professor, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2066383
Record Dates: First submitted 2022-08-15; First posted 2022-08-17 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer Female
Keywords: cancer; metacognition; cognition; Telehealth; activities of daily living
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: After baseline assessment, subjects will be randomized to one of two groups: (1) a 10-session Cognitive Orientation to daily Occupational Performance (CO-OP) intervention; or (2) a 10-session attention control group.
Who Masked: Outcomes Assessor
Masking Description: All outcomes assessors will be blinded to participant study group assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group: Cognitive Orientation to daily Occupational Performance (CO-OP) (Experimental): Each CO-OP session will last 60 minutes and subjects will complete one session per week over the course of 10 weeks. All sessions will be delivered remotely via the Zoom platform.
  Interventions: Behavioral: CO-OP Procedures
- Attention Control Group (Active Comparator): Each session will last 60 minutes and subjects will complete one session per week over the course of 10 weeks. All sessions will be delivered remotely via the Zoom platform.
  Interventions: Behavioral: Attention Control Procedures

INTERVENTIONS:
Behavioral: CO-OP Procedures — CO-OP is a metacognitive strategy training intervention that will be used in this study. First, five functional, everyday life goals are identified collaboratively by the participant and interventionist. In the second meeting, we introduce the approach to the subject and teach the global cognitive strategy (i.e., GOAL-PLAN-DO-CHECK). In all subsequent sessions, this strategy is used as the main problem-solving framework to facilitate skill acquisition.The subject identifies a GOAL, and then is guided by the therapist to discover a PLAN to potentially achieve the goal. The subject is then asked to DO the plan (if feasible during the therapy session otherwise asked to complete at home prior to the next treatment session), and subsequently to CHECK to see if the plan worked, i.e. the goal was achieved. This process is repeated until satisfactory performance is met for each established goal.
  Arms: Treatment Group: Cognitive Orientation to daily Occupational Performance (CO-OP)
Behavioral: Attention Control Procedures — Individuals in the attention control group will have dose-equivalent, weekly virtual contact through the Zoom platform for 12-weeks with a a trained interventionist not involved in CO-OP treatment. The control group will control for interpersonal interaction, maturation effects, and testing effects. The focus of each session will include: (1) social interaction characterized by warmth/empathy and (2) provision of usual care CRCI educational resources (e.g. exercise, using memory aids, minimizing distractions) from MD Anderson Cancer Center. These recommendations will be provided without further instruction. Any questions that arise regarding CRCI the subject is experiencing will be answered. The therapist will debrief with the subject on any changes in CRCI symptoms. The content and duration of each call will be tracked. Each session will be recorded with two randomly selected and reviewed for fidelity.
  Arms: Attention Control Group

SUMMARY:
The first aim of this study is to determine the feasibility of delivering CO-OP remotely to breast cancer survivors, who self-report cancer-related cognitive impairment (CRCI), in preparation for a future R01 trial. The second aim of this study is to assess the effect of CO-OP on activity performance, subjective and objective cognition, and quality of life in a sample of breast cancer survivors who self-report CRCI. The research team hypothesizes that effect size estimations will indicate that CO-OP will have a greater positive effect, compared to attention control, on activity performance, subjective and objective cognition, and quality of life in a sample of breast cancer survivors who self-report CRCI.

DETAILED DESCRIPTION:
Breast cancer survivors often self-report cognitive changes after treatment for cancer (e.g. cancer-related cognitive impairment (CRCI)). These cognitive changes have a devastating impact on everyday life activities, such as work/productivity, community involvement, driving, and financial management. While CRCI would likely be amenable to rehabilitation services, breast cancer survivors face two primary barriers to adequate rehabilitation, including (1) inadequate access to rehabilitation services, and (2) limited effective interventions to address CRCI.

Breast cancer survivors have inadequate access to rehabilitation services to address CRCI. A recent report sponsored by the National Cancer Institute (NCI) concluded that most NCI-designated cancer centers do not have integrated cancer rehabilitation services. Even if comprehensive rehabilitation services were provided by these centers, millions of cancer survivors live in rural areas outside close proximity to a cancer center and are more likely to experience poorer outcomes compared to urban counterparts. If rehabilitation services were provided, proximity to facilities may be a limiting factor in individuals from rural communities receiving rehabilitative care. Access to services has been further curtailed amid the COVID-19 pandemic, with calls building from national organizations for improvements in remote delivery of services.

Metacognitive strategy training (MCST) is a practice standard to address cognitive impairment in other conditions, such as traumatic brain injury and stroke. The Cognitive-Orientation to daily Occupational Performance (CO-OP) approach is a MCST intervention in which subjects are taught a general cognitive strategy that can be applied in known and novel contexts to devise task specific strategies to engage in an activity. The investigators' preliminary data suggest that CO-OP may have a positive impact on activity performance, subjective and objective cognition, and quality of life in breast cancer survivors with CRCI. While current evidence supports the remote delivery of strategy-based interventions like CO-OP, this intervention has not been evaluated in breast cancer survivors with CRCI.

The investigators' overall research hypothesis is that CO-OP can feasibly be administered remotely and will improve activity performance, subjective and objective cognition, and subjective quality of life in breast cancer survivors with CRCI.

ELIGIBILITY:
Inclusion Criteria:

* self-reported CRCI (Cognitive Failures Questionnaire (CFQ) score >30)
* completed full course of chemotherapy at least 6 months, but no later than 3 years, prior to participation
* able to read, write, and speak English fluently
* able to provide valid informed consent
* have a life expectancy of greater than 6 months at time of enrollment
* diagnosed with breast cancer (invasive ductal or lobular BrCA Stages I, II, or III) and completed chemotherapy within the preceding three years
* on stable doses of medications (i.e., no changes in past 60 days)

Exclusion Criteria:

* prior cancer diagnoses of other sites with evidence of active disease within the past year
* active diagnoses of any acute or chronic brain-related neurological conditions that can alter normal brain function (e.g., Parkinson's disease, dementia, cerebral infarcts, traumatic brain injury)
* severe depressive symptoms (Personal Health Questionnaire (PHQ-9) score of ≥21)

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-10-11 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anna E Boone, PhD, OTR/L, Principal Investigator — University of Missouri Occupational Therapy
Locations (1):
- University of Missouri Occupational Therapy Department, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hutchinson AD, Hosking JR, Kichenadasse G, Mattiske JK, Wilson C. Objective and subjective cognitive impairment following chemotherapy for cancer: a systematic review. Cancer Treat Rev. 2012 Nov;38(7):926-34. doi: 10.1016/j.ctrv.2012.05.002. Epub 2012 Jun 2. PMID 22658913
- [Background] O'Farrell E, MacKenzie J, Collins B. Clearing the air: a review of our current understanding of "chemo fog". Curr Oncol Rep. 2013 Jun;15(3):260-9. doi: 10.1007/s11912-013-0307-7. PMID 23483375
- [Background] Reid-Arndt SA, Hsieh C, Perry MC. Neuropsychological functioning and quality of life during the first year after completing chemotherapy for breast cancer. Psychooncology. 2010 May;19(5):535-44. doi: 10.1002/pon.1581. PMID 19472296
- [Background] Reid-Arndt SA, Yee A, Perry MC, Hsieh C. Cognitive and psychological factors associated with early posttreatment functional outcomes in breast cancer survivors. J Psychosoc Oncol. 2009;27(4):415-34. doi: 10.1080/07347330903183117. PMID 19813133
- [Background] Cicerone KD, Dahlberg C, Kalmar K, Langenbahn DM, Malec JF, Bergquist TF, Felicetti T, Giacino JT, Harley JP, Harrington DE, Herzog J, Kneipp S, Laatsch L, Morse PA. Evidence-based cognitive rehabilitation: recommendations for clinical practice. Arch Phys Med Rehabil. 2000 Dec;81(12):1596-615. doi: 10.1053/apmr.2000.19240. PMID 11128897
- [Background] Cicerone KD, Langenbahn DM, Braden C, Malec JF, Kalmar K, Fraas M, Felicetti T, Laatsch L, Harley JP, Bergquist T, Azulay J, Cantor J, Ashman T. Evidence-based cognitive rehabilitation: updated review of the literature from 2003 through 2008. Arch Phys Med Rehabil. 2011 Apr;92(4):519-30. doi: 10.1016/j.apmr.2010.11.015. PMID 21440699
- [Background] Haskins E. Cognitive Rehabilitation Manual: Translating Evidence-Based Recommendations into Practice. Vol 1. Reston, VA: American Congress of Rehabilitation Medicine; 2012.
- [Background] Wolf TJ, Doherty M, Kallogjeri D, Coalson RS, Nicklaus J, Ma CX, Schlaggar BL, Piccirillo J. The Feasibility of Using Metacognitive Strategy Training to Improve Cognitive Performance and Neural Connectivity in Women with Chemotherapy-Induced Cognitive Impairment. Oncology. 2016;91(3):143-52. doi: 10.1159/000447744. Epub 2016 Jul 23. PMID 27449501

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of the recruitment period: September 2022-December 2023
  Types of recruitment: Local cancer registry, cancer support groups, newsletters, social media posts (Facebook, Instagram, Twitter), flyers in the community.
Pre-assignment Details: One participant was enrolled and signed written consent but withdrew during baseline assessment. Therefore, this participant was never randomized.
Period: Overall Study
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Started | 23 | 22
Completed | 21 | 21
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Row population differs from overall due to attrition.
  years | 52.8 (9.7) | 56.5 (10.6) | 53.9 (10.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Row population differs from overall population due to attrition.
  Participants
    Female | 21 | 21 | 42
    Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Row population differs from overall population due to attrition.
  Participants
    Hispanic or Latino | 2 | 0 | 2
    Not Hispanic or Latino | 19 | 21 | 40
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Row population differs from overall population due to attrition.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 0 | 3 | 3
    White | 20 | 17 | 37
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants] — Population: Row population differs from overall population due to attrition.
  participants
    United States | 21 | 21 | 42
Education [Mean (Standard Deviation); unit: years] — Population: Row population differs from overall population due to attrition.
  years | 15.9 (2.4) | 16.0 (2.7) | 15.9 (2.5)
Breast cancer stage [Count of Participants; unit: Participants] — Population: Row population differs from overall population due to attrition.
  Participants
    Invasive Ductal Stage 1 | 6 | 8 | 14
    Invasive Ductal Stage 2 | 5 | 7 | 12
    Invasive Ductal Stage 3 | 6 | 4 | 10
    Invasive Lobular Stage 1 | 2 | 0 | 2
    Invasive Lobular Stage 2 | 1 | 1 | 2
    Invasive Lobular Stage 3 | 1 | 1 | 2
Chemotherapy length [Mean (Standard Deviation); unit: months] — Population: Row population differs from overall population due to attrition.
  months | 5.9 (4.6) | 6.4 (4.3) | 6.2 (4.4)
Time post chemotherapy [Mean (Standard Deviation); unit: months] — Population: Row population differs from overall population due to attrition.
  months | 19.6 (8.9) | 22.9 (9.8) | 21.2 (9.4)
Radiation [Count of Participants; unit: Participants] — Received radiation=yes Did not receive radiation=no Population: Row population differs from the overall population due to attrition.
  Participants
    Yes | 11 | 13 | 24
    No | 10 | 8 | 18
Hormonal therapies [Count of Participants; unit: Participants] — Received hormonal therapies=yes Did not receive hormonal therapies=no Population: Row population differs from overall population due to attrition.
  Participants
    Yes | 15 | 15 | 30
    No | 6 | 6 | 12

OUTCOME MEASURES:

1. Primary Outcome: Telehealth Usability Questionnaire (TUQ)
Description: Measure of telehealth usability from participant's perspective. Specifically, the TUQ measures usefulness and utility of technologies including usefulness, ease of use, effectiveness, reliability, and satisfaction. The TUQ uses a self-report Likert scale of 1 (disagree) to 7 (agree).
Time Frame: After study completion, an average of 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
units on a scale | 6.38 (0.61) | 6.31 (0.61)

2. Primary Outcome: Acceptability of Intervention Measure (AIM)
Description: Measure of intervention acceptability. Self-report Likert scale of 1 (completely disagree) to 5 (completely agree)
Time Frame: After study completion, an average of 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
units on a scale | 4.58 (0.55) | 4.25 (0.58)

3. Primary Outcome: Intervention Appropriateness Measure (IAM)
Description: Measure of intervention appropriateness. Self-report Likert scale of 1 (completely disagree) to 5 (completely agree)
Time Frame: After study completion, an average of 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
units on a scale | 4.43 (0.62) | 3.83 (0.90)

4. Primary Outcome: Feasibility of Intervention Measure (FIM)
Description: Measure of intervention feasibility. Self-report Likert scale of 1 (completely disagree) to 5 (completely agree)
Time Frame: After study completion, an average of 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
units on a scale | 4.64 (0.53) | 4.20 (1.06)

5. Primary Outcome: Canadian Occupational Performance Measure (COPM) Trained Goal Performance
Description: Self-report measure of activity performance. Minimum = 1, Maximum = 10. Higher scores mean better performance.
Time Frame: Pre-intervention (week 0) and post-intervention (week 14)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
units on a scale
  Baseline | 4.4 (1.3) | 4.1 (1.6)
  Post | 6.83 (1.2) | 5.7 (1.7)
Statistical Analysis 1: Comparison: Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) vs Attention Control Group; Test type: Other; Cohen's d effect size = .44, 95% CI 2-sided [-.16 to 1.05]

6. Primary Outcome: NeuroQoL Cognitive Function Short Form
Description: Self-report measure of cognitive ability in daily life activity. Maximum = 5 (never), Minimum = 1 (Very often/several times per day). The total raw score range is 8-40. The t-score is reported with a mean of 50 and standard deviation of 10. Higher scores mean fewer perceived cognitive challenges.
Time Frame: Pre-intervention (week 0) and post-intervention (week 14)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
units on a scale
  Baseline | 36.4 (5.9) | 37.2 (6.3)
  Post | 44.0 (6.8) | 42.6 (6.3)
Statistical Analysis 1: Comparison: Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) vs Attention Control Group; Test type: Other; Cohen's d effect size = .42, 95% CI 2-sided [-.19 to 1.03]

7. Primary Outcome: Canadian Occupational Performance Measure (COPM) Trained Goal Satisfaction
Description: Self-report measure of satisfaction level with activity performance. Minimum = 1, Maximum = 10. Higher scores mean higher satisfaction.
Time Frame: After study completion, an average of 14 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
units on a scale
  Baseline | 4.2 (2.3) | 3.4 (1.8)
  Post | 6.9 (1.5) | 5.4 (2.3)
Statistical Analysis 1: Comparison: Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) vs Attention Control Group; Test type: Other; Cohen's d effect size = .31, 95% CI 2-sided [-.30 to 0.93]

8. Secondary Outcome: Functional Assessment of Cancer Therapy-Breast (FACT-B)
Description: Self-report measure of quality of life for breast cancer survivors. Domains include questions related to physical, emotional, social, and functional well-being, as well as additional concerns. Minimum = 0 (not at all), Maximum = 4 (very much). The range of scores is 0 to 148. Higher scores indicate decreased perceived well-being and quality of life.
Time Frame: Pre-intervention (week 0) and post-intervention (week 14)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
units on a scale
  Baseline | 91.9 (23.3) | 90 (21.6)
  Post | 99.8 (21.8) | 104.3 (14.3)
Statistical Analysis 1: Comparison: Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) vs Attention Control Group; Test type: Other; Cohen's d effect size = -.42, 96% CI 2-sided [-1.04 to 0.21]

9. Secondary Outcome: Delis-Kaplan Executive Function System (DKEFS)- Color-Word Interference Subtest
Description: Objective measure of inhibition and cognitive flexibility. Data are presented for condition 4 of Number/Letter switching. Age-adjusted scale scores with a mean of 10 and standard deviation of 3 are reported. The total range of scores is 1-19. Higher scores indicate better performance.
Time Frame: Pre-intervention (week 0) and post-intervention (week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 10.2 (2.5) | 9.9 (2.4)
  Post | 11.2 (3.1) | 10.3 (2.6)

10. Secondary Outcome: Wechsler Adult Intelligence Scale (WAIS)-IV Letter-Number, Coding, Symbol Search Subtest
Description: Objective measure of cognitive performance. The Letter-Number subtest measures working memory. The Coding and Symbol Search subtest measure processing speed. Higher scores indicate better cognitive performance. Age adjusted scaled scores with a mean of 10 and standard deviation of 3 are reported. Range of reported scores is 1 to 19.
Time Frame: Pre-intervention (week 0) and post-intervention (week 14)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
score on a scale
  Letter Number Baseline | 9.4 (2.4) | 9.6 (3.6)
  Letter Number Post | 10.6 (3.1) | 10.1 (2.3)
  Symbol Search Baseline | 10.5 (2.6) | 9.2 (2.3)
  Symbol Search Post | 12.2 (2.3) | 11.1 (3.1)
  Coding Baseline | 10.6 (2.6) | 9.8 (2.6)
  Coding Post | 9.4 (2.7) | 9.8 (2.6)

11. Secondary Outcome: Brief Visuospatial Memory Test -Revised Trial 1
Description: Objective measure of episodic memory. Participant is presented with six geometric figures for 10 seconds on three different occasions, and then asked to draw the six figures on a separate sheet of paper in the correct order. Increased errors may indicate challenges with episodic memory. T-scores are reported with a mean of 50 and standard deviation of 10. Higher scores indicate better performance.
Time Frame: Pre-intervention (week 0) and post-intervention (week 14)
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
T-score
  Baseline | 51.0 (11.4) | 56.4 (12.0)
  Post | 47.0 (9.4) | 54.8 (16.2)

12. Secondary Outcome: Paced Auditory Serial Addition Test
Description: Objective measure of working memory. Participant is presented with single digits every 2 seconds and asked to add each digit to the one immediately prior to it. Total score is out of 60 points, with increased errors indicating challenges with working memory.
Time Frame: Pre-intervention (week 0) and post-intervention (week 14)
Measure: Mean (Standard Deviation); unit: number correct
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
number correct
  Baseline | 26.8 (10.2) | 26.2 (6.8)
  Post | 29.9 (10.7) | 25.7 (9.4)

13. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Ability to Participate in Social Roles and Activities
Description: Self-report measure of ability to participate in social roles and activities. Higher scores reflect higher abilities. T-scores are reported with a mean of 50 and a standard deviation of 10.
Time Frame: Pre-intervention (week 0) and post-intervention (week 14)
Population: T-scores are used with mean of 50 and standard deviation of 10
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
Number analyzed (Participants) | 21 | 21
T-score
  Baseline | 45.5 (8.5) | 47.1 (9.7)
  Post | 48.2 (9.7) | 49.7 (6.7)
Statistical Analysis 1: Comparison: Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) vs Attention Control Group; Test type: Other; Cohen's d effect size = 0.01, 95% CI 2-sided [-.61 to .64]

ADVERSE EVENTS:
Time Frame: Through study completion, up to 14 weeks
Arm/Group | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) | Attention Control Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 3/23 | 0/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group: Cognitive Orientation to Daily Occupational Performance (CO-OP) (N=23) | Attention Control Group (N=22)
Fall in community (Injury, poisoning and procedural complications) | 1 (1) | 0 — Pt was walking in the community when she tripped and fell, resulting in R humeral neck fracture. Pt's husband was present and accompanied her to the physician. She received a sling for RUE. Pt's schedule was revised to accommodate all 10 sessions.
Fall at home (Injury, poisoning and procedural complications) | 1 (2) | 0 — Pt reported that she fell due to tripping 2x at home (same day). She had no injuries besides soreness and no medical attention was required. Pt's husband was present. No disruption to treatment schedule.
Bleeding at incision site (Injury, poisoning and procedural complications) | 1 (1) | 0 — Pt had medical procedure on Monday 9/11/23 and on Friday 9/15/23 had bleeding at incision site. Pt went to ER for treatment and rested over the weekend. Pt returned to work on Monday 9/18/23 and did not miss any study sessions as a result.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/45/NCT05505045/Prot_SAP_ICF_000.pdf